CLINICAL TRIAL: NCT06071247
Title: Application and Translational Research of 3D Printed Models in the Surgical Treatment of Common Bile Duct Stones Under Endoscopic Retrograde Cholangiopancreatography
Brief Title: Application and Translational Research of 3D Printed in Treatment of Choledocholithiasis Under ERCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiawei Qin (Other)
Responsible Party: Sponsor-Investigator, Jiawei Qin, Resident physician, Guangdong Second Provincial General Hospital
Organization: Guangdong Second Provincial General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D-A2020005
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Common Bile Duct Calculi
Keywords: Common Bile Duct Calculi ;ERCP ;3D printed models
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use 3D printed models group (Experimental): This group will use 3D printed models for preoperative simulation planning and then undergo surgery
  Interventions: Other: 3D printed models
- Not use 3D printed models group (No Intervention): This group will undergo surgery directly without using 3D printed models.

INTERVENTIONS:
Other: 3D printed models — 3D printed simulation models of the stomach, duodenum, common bile duct, and pancreatic duct structures using a combination of soft and hard materials
  Arms: Use 3D printed models group

SUMMARY:
The goal of this clinical trial is to learn about Application and translational research of 3D printed models in the surgical treatment of common bile duct stones under endoscopic retrograde cholangiopancreatography. The main question it aims to answer are:Compare the differences in stone removal time, surgical complications, and surgical success rate during ERCP (+EST) surgery between 30 patients who used 3D printing preoperative simulation and 30 patients who did not use it.

Participating patients will be divided into two groups, one group of 30 patients will use 3D printed models for preoperative simulation planning and then undergo surgery, and the other group will undergo surgery directly without using 3D printed models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple or single common bile duct stones (total stone diameter ≤1.5 cm)
* Patients who voluntarily participated in the study and signed the consent form

Exclusion Criteria:

* Patients with various underlying diseases, such as diabetes, coronary heart disease, and hypertension, that would increase the risk of surgery and affect the outcome of surgery
* Patients who have had cholangiojejunostomy or Roux-en-Y anastomosis
* Combined with intrahepatic bile duct stones require surgical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
operation time | intraoperatively
  The operation time of the 3D printed model group was shorter than that of the control group
Surgery success rate | intraoperatively
  The surgery success rate of the 3D printed model group was higher than that of the control group
amount of bleeding | intraoperatively
  The amount of bleeding of the 3D printed model group was lower than that of the control group
complications | Within 3 days to 1 month after surgery
  The complications of the 3D printed model group was lower than that of the control group

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Li, Principal Investigator — Guangdong Second Provincial General Hospital